CLINICAL TRIAL: NCT01278160
Title: An Extension Trial of BIAsp-3756, Explorative Comparison of Biphasic Insulin Aspart 30 Twice Daily With Two Different Initial Dosage Split Regimens on the Effect of Glycaemic Control in Chinese Type 2 Diabetes Patients
Brief Title: Comparison of Biphasic Insulin Aspart 30 Twice Daily With Two Different Initial Dosage Split Regimens in Subjects With Type 2 Diabetes: An Extension to Trial BIASP-3756
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-3883; U1111-1118-0330 (Other: WHO)
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Results first posted 2012-10-18 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIAsp 30 (2:1) (Experimental): After discontinuation of previous treatment of once daily biphasic insulin aspart 30 (BIAsp 30) or insulin glargine combined with metformin and glimepiride in trial BIAsp-3756, subjects were adminstered BIAsp 30 twice daily with initial dosage split regimen of 2/3 and 1/3 total daily dose before breakfast and before dinner, respectively combined with metformin administered orally with meals
  Interventions: Drug: biphasic insulin aspart 30; Drug: metformin
- BIAsp 30 (1:1) (Experimental): After discontinuation of previous treatment of once daily biphasic insulin aspart 30 (BIAsp 30) or insulin glargine combined with metformin and glimepiride in trial BIAsp-3756, subjects were adminstered BIAsp 30 twice daily with initial dosage split regimen of 1/2 and 1/2 total daily dose before breakfast and before dinner, respectively combined with metformin administered orally with meals
  Interventions: Drug: biphasic insulin aspart 30; Drug: metformin

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Administered subcutaneously (under the skin), twice daily with a dosage of 2/3 and 1/3 total daily dose before breakfast and before dinner, in combination with metformin.
  Arms: BIAsp 30 (2:1)
Drug: biphasic insulin aspart 30 — Administered subcutaneously (under the skin), twice daily with a split dosage of 1/2 and 1/2 total daily dose before breakfast and before dinner, in combination with metformin.
  Arms: BIAsp 30 (1:1)
Drug: metformin — Tablets 500 mg administered orally with meals. Pre-trial dose and regimen unchanged

SUMMARY:
This trial is conducted in Asia. The aim of the trial is to compare the effect on glycaemic control of biphasic insulin aspart 30 twice daily with two different dosage split regimens for Chinese subjects with type 2 diabetes who did not achieve the treatment target of a glycosylated haemoglobin A1c (HbA1c) below 7% in trial BIASP-3756 (NCT01123980).

ELIGIBILITY:
Inclusion Criteria:

* Finalised 24 weeks of treatment with once daily BIAsp 30 or insulin glargine in combination with metformin and glimepiride in trial BIAsp-3756
* HbA1c above or equal to 7.0%
* Body Mass Index (BMI) below or equal to 40.0 kg/m2

Exclusion Criteria:

* Known hypoglycaemia unawareness or recurrent major hypoglycaemic episodes in trial BIAsp-3756
* Known proliferative retinopathy or maculopathy requiring acute treatment
* Any disease or condition which the Investigator (trial physician) feels would interfere with the trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Beijing, Beijing Municipality, China

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 20 sites in China.
Pre-assignment Details: All subjects who completed the 24 week treatment and did not achieve the target of glycosylated haemoglobin A1c (HbA1c) below 7% in trial BIAsp-3756 (NCT01123980) were offered the possibility to go into BIAsp-3883. Subjects continued their previous treatment unchanged from trial BIASP-3756 and throughout the one-week screening period.
Period: Overall Study
Arm/Group | BIAsp 30 (2:1) | BIAsp 30 (1:1)
Started | 89 | 90
Completed | 84 | 84
Not Completed | 5 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Unclassified | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIAsp 30 (2:1) | BIAsp 30 (1:1) | Total
Number analyzed (Participants) | 89 | 90 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (9.9) | 57.1 (9.4) | 56.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 48 | 95
  Male | 42 | 42 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 89 | 90 | 179
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 89 | 90 | 179
Height [Mean (Standard Deviation); unit: cm] | 165.2 (7.4) | 165.3 (8.4) | 165.3 (7.9)
Weight [Mean (Standard Deviation); unit: kg] | 72.2 (11.1) | 72.3 (11.6) | 72.2 (11.3)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.40 (3.44) | 26.36 (3.28) | 26.38 (3.35)
Glycosylated haemoglobin (HbA1c) at screening [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 7.80 (0.65) | 7.80 (0.73) | 7.80 (0.69)
Duration of diabetes [Mean (Standard Deviation); unit: years] — Number of years since diagnosis
  years | 9.08 (6.05) | 10.23 (5.89) | 9.65 (5.98)
Diabetic complications [Number; unit: participants]
  Yes | 16 | 22 | 38
  No | 69 | 67 | 136
  Missing data | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin A1c (HbA1c) From Baseline
Time Frame: Week 0, week 16
Population: Full analysis set using LOCF (last observation carried forward) consists of all randomised subjects who were exposed to at least one dose of the trial product(s). Six patients discontinued trial without any post randomisation HbA1c measurements.
Measure: Least Squares Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | BIAsp 30 (2:1) | BIAsp 30 (1:1)
Number analyzed (Participants) | 86 | 87
percentage of glycosylated haemoglobin | -0.13 (0.08) | -0.12 (0.08)
Statistical Analysis 1: Comparison: BIAsp 30 (2:1) vs BIAsp 30 (1:1); The null hypothesis is H0: μBIAsp 30 (2:1) - μBIAsp 30 (1:1) = 0 against the alternative hypothesis HA: μBIAsp 30 (2:1) - μBIAsp 30 (1:1) ≠ 0. This trial is an extension to BIAsp-3756 (NCT01123980), hence no particular sample size calculation was made; Test type: Superiority or Other; ANCOVA; The estimates were from a normal linear regression model with treatment and previous insulin as factors, and baseline value as a covariate; Mean Difference (Net) = -0.01, 95% CI [-0.24 to 0.22], Standard Error of Mean 0.12

2. Secondary Outcome: 9-point SMPG (Self Measured Plasma Glucose) Profile
Description: A 9-point SMPG profile included measurements before and 120 minutes after start of breakfast, lunch and main evening meal, measurements prior to bedtime and at 2:00 -4:00 a.m., and one before breakfast the following day
Time Frame: Week 16
Population: Full analysis set using LOCF (last observation carried forward) consists of all randomised subjects who were exposed to at least one dose of the trial product(s).
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BIAsp 30 (2:1) | BIAsp 30 (1:1)
Number analyzed (Participants) | 89 | 90
mmol/L
  Before breakfast | 6.02 (1.09) | 6.23 (1.23)
  2 hours after breakfast | 8.56 (2.28) | 8.61 (2.41)
  Before lunch | 6.42 (1.62) | 6.79 (2.49)
  2 hours after lunch | 8.91 (2.59) | 9.17 (2.70)
  Before dinner | 6.64 (1.95) | 7.07 (2.07)
  2 hours after dinner | 7.92 (2.34) | 7.94 (1.98)
  Bedtime | 7.29 (1.99) | 7.03 (1.91)
  2:00 - 4:00 a.m. | 6.05 (1.53) | 6.34 (1.65)
  Before breakfast the following day | 6.30 (1.38) | 6.22 (1.40)
Statistical Analysis 1: Comparison: BIAsp 30 (2:1) vs BIAsp 30 (1:1); A mixed effect model was fitted to the 9-point SMPG profile data. The model included treatment, time, interaction between treatment and time and previous therapy (BIAsp 30 OD/insulin glargine OD) as factors and subject as random effect. From the model, mean profile by treatment and relevant treatment differences was estimated and explored; Test type: Superiority or Other; p = 0.2569, Mixed Models Analysis — P-value for parallelism was overall test for parallel time profiles between treatment groups, i.e. time by treatment group interaction effect; Mixed models analysis = 0.20, 95% CI [-0.15 to 0.56] — Confidence interval is before breakfast profile
Statistical Analysis 2: Comparison: BIAsp 30 (2:1) vs BIAsp 30 (1:1); A mixed effect model was fitted to the 9-point SMPG profile data. The model included treatment, time, interaction between treatment and time and previous therapy (BIAsp-30 once daily (OD)/insulin glargine OD) as factors and subject as random effect. From the model, mean profile by treatment and relevant treatment differences was estimated and explored; Test type: Superiority or Other; p = 0.8120, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mixed models analysis = 0.09, 95% CI [-0.63 to 0.80] — Confidence interval is two hours after breakfast profile
Statistical Analysis 3: Comparison: BIAsp 30 (2:1) vs BIAsp 30 (1:1); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.2843, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mixed model analysis = 0.35, 95% CI [-0.29 to 0.99] — Confidence interval is before lunch profile
Statistical Analysis 4: Comparison: BIAsp 30 (2:1) vs BIAsp 30 (1:1); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.4614, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mixed model analysis = 0.30, 95% CI [-0.50 to 1.11] — Confidence interval is two hours after lunch profile
Statistical Analysis 5: Comparison: BIAsp 30 (2:1) vs BIAsp 30 (1:1); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.1591, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mixed model analysis = 0.44, 95% CI [-0.17 to 1.04] — Confidence interval is before dinner profile
Statistical Analysis 6: Comparison: BIAsp 30 (2:1) vs BIAsp 30 (1:1); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.9327, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mixed model analysis = 0.03, 95% CI [-0.63 to 0.69] — Confidence interval is two hours after dinner profile
Statistical Analysis 7: Comparison: BIAsp 30 (2:1) vs BIAsp 30 (1:1); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.4063, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mixed model analysis = -0.25, 95% CI [-0.84 to 0.34] — Confidence interval is bedtime profile
Statistical Analysis 8: Comparison: BIAsp 30 (2:1) vs BIAsp 30 (1:1); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.2198, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mixed model analysis = 0.30, 95% CI [-0.18 to 0.79] — Confidence interval is 2.00 - 4.00 a.m. profile
Statistical Analysis 9: Comparison: BIAsp 30 (2:1) vs BIAsp 30 (1:1); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.8424, Mixed Models Analysis; Mixed model analysis = -0.04, 95% CI [-0.47 to 0.38] — Confidence interval is before breakfast the following day profile

3. Secondary Outcome: Percentage of Subjects Achieving HbA1c Below 7.0%
Description: The percentage of subjects achieving the treatment target for glycosylated haemoglobin A1c (HbA1c) after 16 weeks of treatment
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | BIAsp 30 (2:1) | BIAsp 30 (1:1)
Number analyzed (Participants) | 89 | 90
percentage of subjects | 12.4 | 14.4
Statistical Analysis 1: Comparison: BIAsp 30 (2:1) vs BIAsp 30 (1:1); Responder analyses were based on logistics regression model using treatment and previous therapy (BIAsp 30 OD or insulin glargine OD) as factors and baseline HbA1c as covariate; Test type: Superiority or Other; p = 0.7312, Regression, Logistic; Odds Ratio (OR) = 0.86, 95% CI [0.36 to 2.06] — The odds ratio and 95% confidence interval for the HbA1c below 7% treatment target were included

4. Secondary Outcome: Percentage of Subjects Achieving HbA1c Below or Equal to 6.5%
Description: as for outcome 3
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | BIAsp 30 (2:1) | BIAsp 30 (1:1)
Number analyzed (Participants) | 89 | 90
percentage of subjects | 2.2 | 7.8
Statistical Analysis 1: Comparison: BIAsp 30 (2:1) vs BIAsp 30 (1:1); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.1257, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.27, 95% CI [0.05 to 1.44] — The odds ratio and 95% confidence interval for the HbA1c below or equal to 6.5% treatment target were included

5. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes
Description: Treatment emergent hypoglycaemic episodes (hypos): those that happened between treatment and one day after last drug day. Hypos summarised based on American Diabetes Association classification. Severe hypos: episodes requiring another person to actively administer resuscitative actions. Minor hypos: episodes with symptoms with plasma glucose below 3.1 mmol/L (56 mg/dL) handled by the subject, or any asymptomatic plasma glucose below 3.1 mmol/L (56 mg/dL). Diurnal period: between 06:00 and 23:59 (both included). Nocturnal period: between 00:00 and 05:59 a.m. (both included).
Time Frame: Weeks 0-16
Population: as for outcome 2
Measure: Number; unit: episodes
Arm/Group | BIAsp 30 (2:1) | BIAsp 30 (1:1)
Number analyzed (Participants) | 89 | 90
episodes
  All episodes | 108 | 143
  Nocturnal | 18 | 11
  Diurnal | 84 | 127
  Severe | 0 | 0
  Minor | 20 | 35
Statistical Analysis 1: Comparison: BIAsp 30 (2:1) vs BIAsp 30 (1:1); The number of hypos was analysed using a negative binomial regression model with a log-link function and the logarithm of the time period in which a hypo is considered emergent as offset. The model included treatment and previous therapy (BIAsp 30 OD/insulin glargine OD) as factors. The rate ratio was estimated and 95% confidence intervals were calculated accordingly; Test type: Superiority or Other; p = 0.1911, Negative binomial regression model; Rate ratio = 0.72, 95% CI [0.43 to 1.18] — For all episodes
Statistical Analysis 2: Comparison: BIAsp 30 (2:1) vs BIAsp 30 (1:1); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.2949, Negative binomial regression model; Rate ratio = 1.61, 95% CI [0.66 to 3.92] — For nocturnal episodes
Statistical Analysis 3: Comparison: BIAsp 30 (2:1) vs BIAsp 30 (1:1); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0770, Negative binomial regression model; Rate ratio = 0.63, 95% CI [0.38 to 1.05] — For diurnal episodes
Statistical Analysis 4: Comparison: BIAsp 30 (2:1) vs BIAsp 30 (1:1); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.1687, Negative binomial regression model; Rate ratio = 0.56, 95% CI [0.25 to 1.27] — For minor episodes

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a timespan of 17 weeks.
Description: The safety analysis set contained all subjects exposed to at least one dose of investigational products.
Arm/Group | BIAsp 30 (2:1) | BIAsp 30 (1:1)
Serious Adverse Events (participants affected / at risk) | 1/89 | 2/90
Other Adverse Events (participants affected / at risk) | 0/89 | 0/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIAsp 30 (2:1) (N=89) | BIAsp 30 (1:1) (N=90)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right to not release data until specified milestones, e.g. when the clinical trial report is available. At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.